CLINICAL TRIAL: NCT00183729
Title: Memantine for Enhancement of Rehabilitation Efficacy and Prevention of Major Depressive Disorder in Older Adults
Brief Title: Memantine Treatment for Improving Rehabilitation Outcomes and Preventing Depression in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric Lenze (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Eric Lenze, Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23MH064196-02 (NIH); K23MH064196-02 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Depression
Keywords: Major depressive disorder; Rehabilitating; Elderly; Apathy
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Lethargy | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (1) (Experimental): Memantine for 12 weeks
  Interventions: Drug: Memantine
- Placebo (2) (Placebo Comparator): Placebo for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine dosage is started at 10 mg daily and is increased at Week 1 as tolerated to 10 mg two times a day.
  Other Names: Namenda
  Arms: Memantine (1)
Other: Placebo — Placebo distribution is planned to mimic the active drug.
  Arms: Placebo (2)

SUMMARY:
This study will evaluate the effectiveness of memantine in improving rehabilitation outcomes and preventing major depressive disorder in older adults who have been admitted to a rehabilitation hospital for a hip fracture or cardiopulmonary condition.

DETAILED DESCRIPTION:
Depression is a serious medical illness that is often difficult to diagnose and treat. It occurs in people of all ages, but is often overlooked in older adults. Depression frequently co-occurs with other serious illnesses, and may be mistaken by both patients and health care givers as a normal consequence of the illness. However, these misconceptions toward depression contribute to the underdiagnosis and undertreatment of depressive disorders in older people. In turn, depression may hinder a patient's recovery from an illness. This study will evaluate the effectiveness of memantine in improving rehabilitation outcomes and preventing major depressive disorder in older adults who have been admitted to a rehabilitation hospital for a hip fracture or a cardiopulmonary condition.

This double-blind study will last for 12 months. Participants will be randomly assigned to receive either placebo or memantine, which is a drug that is often used to treat Alzheimer's disease. Both memantine and placebo will be administered to participants for 12 weeks. All participants will be followed for an additional 40 weeks. Outcome measurements will include participants' depressive symptoms, motivation, and learned helplessness. In addition, medication side effects, functional outcome, and incidence of major depressive disorder will be measured. All measurements will be taken at Week 12 and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a skilled nursing facility for rehabilitation within 3 months of recent disabling medical event (e.g., hip fracture)
* Medically stable (e.g., no active seizures, delirium, unstable pulse/blood pressure)

Exclusion Criteria:

* Aphasia or cognitive impairments sufficiently severe to prevent valid assessment (e.g., a score of less than 22 on the Mini Mental State Examination)
* Current major depressive episode
* History of or current psychosis or mania
* Current substance or alcohol abuse or dependence (within 3 months of study entry)
* Current use of memantine
* Sensitivity or contraindication to memantine
* End-stage kidney, liver, heart, or lung disease
* Recent hemorrhagic stroke
* A FIM score of greater than 70 (on a 91 point scale)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
study has small sample size and is unlikely to be useful for data sharing efforts; however, interested researchers can contact the first author via email.

REFERENCES:
- [Result] Lenze EJ, Skidmore ER, Begley AE, Newcomer JW, Butters MA, Whyte EM. Memantine for late-life depression and apathy after a disabling medical event: a 12-week, double-blind placebo-controlled pilot study. Int J Geriatr Psychiatry. 2012 Sep;27(9):974-80. doi: 10.1002/gps.2813. Epub 2011 Dec 16. PMID 22173933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects were randomized
Pre-assignment Details: No significant events. Please see Lenze et al, Int J of Geriatric Psychiatry 2012 article for details.
Period: Overall Study
Arm/Group | Memantine (1) | Placebo (2)
Started | 17 | 18
Completed | 14 | 13
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine (1) | Placebo (2) | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.1 (9.7) | 78 (9.2) | 79.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Hamilton depression rating scale ; scale ranges 0 (no symptoms) to 52 (severe depression)
Time Frame: week 0, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine (1) | Placebo (2)
Number analyzed (Participants) | 17 | 18
units on a scale
  Week 0 | 12.5 (3.6) | 13.4 (3.7)
  Week 12 | 7 (1.5) | 5.2 (1.5)
Statistical Analysis 1: Comparison: Memantine (1) vs Placebo (2); Null: the two groups would not differ in depressive symptoms over time (ie both groups would improve equally in terms of their depressive symptoms) Power calculation: none; this was a pilot study; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Final Values) = 2, Standard Error of Mean 2

2. Secondary Outcome: Incidence of Major Depressive Disorder
Description: cumulative incidence over 12 weeks of follow-up
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Memantine (1) | Placebo (2)
Number analyzed (Participants) | 17 | 18
Participants | 3 | 1

3. Secondary Outcome: Functional Recovery
Description: Functional Independence Msure, 13-item motor subscale (scale ranges 13-91, higher scores = better function)
Time Frame: week 0, week 12
Population: intent to treat analysis; data presented are the week 12 data from the mixed effect model
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Memantine (1) | Placebo (2)
Number analyzed (Participants) | 17 | 18
units on a scale | 73 (7) | 81 (6)
Statistical Analysis 1: Comparison: Memantine (1) vs Placebo (2); Null hypothesis: functional recovery would be the same in both groups. Power calculation: none. This was a pilot study; Test type: Superiority — (no comments); p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 8, Standard Error of Mean 7

ADVERSE EVENTS:
Arm/Group | Memantine (1) | Placebo (2)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less